CLINICAL TRIAL: NCT00209768
Title: Randomised, Prospective Study of the Use of In-Line Filtration on the Reduction of Complication Rate in Critically Ill Children
Brief Title: Use of In-Line Filtration in Critically Ill Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Pall Corporation (Other); B. Braun Melsungen AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3702
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-09

CONDITIONS: Critical Illness
Keywords: pediatric intensive care; critically ill children; in-line filtration; prospective randomized study; complications; sepsis; SIRS; thrombosis; organ failure
MeSH Terms: conditions — Critical Illness; Sepsis; Thrombosis

INTERVENTIONS:
Device: Filter: NOE96E, ELD96E, NLF1E, TNA1E

SUMMARY:
The purpose of this study is to determine whether the use of in-line filtration shows any effect on the outcome of sepsis, systemic inflammatory response syndrome (SIRS), thrombosis, or organ failure in critically ill children admitted to the pediatric intensive care unit (PICU).

DETAILED DESCRIPTION:
Scientific background:

Particulate contamination of infusion solutions and their systemic administration during infusion therapy has been linked to various clinical problems.

Organ failure and Multi-Organ Failure (MOV):

It is well established that the pathophysiology of MOV involves deteriorations of the microcirculation and integrity of endothelial cells. As a consequence of this an imbalance between pro- and anticoagulatory factors may develop and microthrombi may form. Mediators like tissue factor (TF) and platelet activating factor (PAF) have been linked to the formation of microthrombi.

Particles have been discussed as a causative agent for this syndrome by various authors. Their effect on morbidity and mortality of patients has however not yet been established.

Particles may have additional harmful effects:

* Direct thrombogenesis by the particle material
* Damaging endothelial cells in the capillary network
* Embolisation of the pulmonary vasculature
* Acting as a cristallisation focus for the development of granuloma
* Promoting the formation of Giant Cells

Various authors have shown that the use of end line infusion filters significantly reduces the rate of thrombophlebitis. A recently published study by van Lingen et al. (2004) also showed that the use of end line infusion filters significantly reduced the rate of overall complications in neonates.

Study Hypothesis:

The use of end line positively charged 0.2 µm and uncharged 1.2 µm infusion filters will prevent particles, microorganisms and their endotoxins from the infusate to enter the patient's circulation in the study group and will reduce significantly the complication rate of these patients.

The following clinical diagnoses are defined as "Complications". They are main contributors to morbidity and mortality in intensive care wards:

* catheter related thrombosis of the central veins
* sepsis with proven infectious organisms
* Septic syndrome without proven infectious organisms
* Failure of one of the following organs/systems

  1. Lung
  2. Kidney
  3. Liver
  4. Circulation

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to pediatric intensive care unit (PICU)

Exclusion Criteria:

* Suspected death within 48 hours
* Duration of PICU stay less than 6 hours
* Patients recruited for Simulect or Sintra Study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 821 (Actual)
Dates: Start 2005-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Sepsis
Thrombosis
SIRS
Organ failure
Composite primary outcome including "sepsis, SIRS, thrombosis, organ failure"

SECONDARY OUTCOMES:
Duration of Pediatric Intensive Care Unit stay
Duration of overall hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sasse, Consultant, Study Director — Medical School Hannover; Thomas Jack, Doctor, Principal Investigator — Medical School Hannover
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Lamping F, Jack T, Rubsamen N, Sasse M, Beerbaum P, Mikolajczyk RT, Boehne M, Karch A. Development and validation of a diagnostic model for early differentiation of sepsis and non-infectious SIRS in critically ill children - a data-driven approach using machine-learning algorithms. BMC Pediatr. 2018 Mar 15;18(1):112. doi: 10.1186/s12887-018-1082-2. PMID 29544449
- [Derived] Boehne M, Jack T, Koditz H, Seidemann K, Schmidt F, Abura M, Bertram H, Sasse M. In-line filtration minimizes organ dysfunction: new aspects from a prospective, randomized, controlled trial. BMC Pediatr. 2013 Feb 6;13:21. doi: 10.1186/1471-2431-13-21. PMID 23384207
- [Derived] Jack T, Boehne M, Brent BE, Hoy L, Koditz H, Wessel A, Sasse M. In-line filtration reduces severe complications and length of stay on pediatric intensive care unit: a prospective, randomized, controlled trial. Intensive Care Med. 2012 Jun;38(6):1008-16. doi: 10.1007/s00134-012-2539-7. Epub 2012 Apr 12. PMID 22527062